CLINICAL TRIAL: NCT03001674
Title: Clinical Hemodynamic Study of Balloon Counterpulsation in Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IABP_Hemodynamics
Record Dates: First submitted 2014-03-27; First posted 2016-12-23 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IABP recipient (Experimental): Referred for clinically indicated right heart catheterization with intervention of IABP placement prior to LVAD surgery.
  Interventions: Device: Conductance catheterization
- Control (Experimental): Control subjects undergoing left heart catheterization with an LV ejection fraction > 50%, and without a history of heart failure symptoms who did not receive IABP therapy were enrolled.
  Interventions: Device: Conductance catheterization

INTERVENTIONS:
Device: Conductance catheterization — CD Leycom Conductance Catheter

SUMMARY:
The primary objective of this study is to develop normative hemodynamic data (means and standard deviations) for the intra-aortic balloon pump (IABP) using pressure-volume loop and 3D-echocardiographic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 18-75 years of age
* NYHA Class III-IV heart failure at the time of MEGA deployment
* Stage C-D systolic heart failure
* Non-ischemic cardiomyopathy
* Preserved right ventricular function defined by 2D-echocardiography
* Clinically indicated left and right heart catheterization and MEGA-IABP placement
* Clinically indicated MEGA-IABP support for 12 hours minimum

Exclusion Criteria:

* Ischemic cardiomyopathy
* Active myocardial ischemia or acute coronary syndrome
* Severe peripheral vascular disease
* Severe aortic or mitral valve insufficiency
* Severe aortic or mitral valve stenosis
* Right ventricular failure
* Inability to tolerate left and right heart catheterization
* Severe hemodynamic instability defined as a systolic BP <80mmHg despite vasopressor/inotropic support
* Sustained ventricular tachycardia (>10 beats) within 24 hours and/or ventricular fibrillation within 24 hours
* Pacemaker dependent rhythm
* Left ventricular thrombus
* Rapid atrial fibrillation (HR>120 bpm)
* Unable to provide informed consent
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Navin Kapur, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients with advanced HF from 2014 to 2015 at Tufts Medical Center referred for clinically indicated RHC and IABP placement prior to LVAD surgery. Five control subjects undergoing left heart catheterization with an LV ejection fraction > 50%, and without a history of heart failure symptoms who did not receive IABP therapy were enrolled.
Groups:
- IABP Recipient: Prospective, double-arm, pilot study.
  Conductance catheterization: CD Leycom Conductance Catheter
- Control Group: Control subjects undergoing left heart catheterization with an LV ejection fraction > 50%, and without a history of heart failure symptoms who did not receive IABP therapy were enrolled.
Period: Overall Study
Arm/Group | IABP Recipient | Control Group
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IABP Recipient | Control | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 54 (13) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.07 (0.33) | 2.22 (0.15) | 2.12 (0.28)

OUTCOME MEASURES:

1. Primary Outcome: Impact of Intra-aortic Balloon Pump Activation on Left Ventricular Stroke Work.
Description: We will be measuring left ventricular stroke work using a conductance catheter before and immediately after activation of an intra-aortic balloon pump (IABP). Left ventricular stroke work is quantified as the product of left ventricular pressure and volume. Conductance catheters are the primary method available for clinical measurement of left ventricular volume and pressure.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mmHg-mL
Arm/Group | IABP Recipient | Control
Number analyzed (Participants) | 10 | 5
mmHg-mL
  Stroke work without IABP | 939 (302) | 5628 (2866)
  Stroke work with IABP | 667 (210) | NA (NA) — Number value for control patients (who did not receive an IABP) should be 'not applicable'

ADVERSE EVENTS:
Arm/Group | IABP Recipient | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

LIMITATIONS AND CAVEATS:
Small number of patients studied. Non-randomized study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No